CLINICAL TRIAL: NCT04942119
Title: Impact of Long-term Serum Magnesium and Potassium Levels Optimization and Multifactorial Adherence Intervention on the Progression of Diabetic Kidney Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: United Arab Emirates University (Other)
Responsible Party: Principal Investigator, Marwan El-Deyarbi, Research Assistant, United Arab Emirates University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SEHA-IRB-021
Record Dates: First submitted 2021-05-21; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Diabetic Kidney Disease; Potassium Imbalance; Magnesium Deficiency
Keywords: Diabetic kidney disease, Magnesium, Potassium, medication adherence, diet adherence, mobile application, fixed medication possession ratio.
MeSH Terms: conditions — Diabetic Nephropathies; Magnesium Deficiency; Medication Adherence

STUDY DESIGN:
Intervention Model Description: A randomized, single-blinded, control study of 160 national UAE citizen patients who have been diagnosed with type 2 diabetes mellitus and will attend the endocrinology or chronic disease clinic (CDC) and having follow-up schedules in an ambulatory healthcare services (AHS) clinic, UAE.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine standard care group (No Intervention): This group will continue to receive the usual recommended care provided in the clinic and usual follow-up appointment as well as clinical assessment. Any required nutrition education by the dietitian or medication counseling will be provided at any visit or when requested.
- Multifactorial intervention group (Experimental): 1. Correction of magnesium and/or potassium levels, and correction of the underlying disease, if possible by a endocrinologist.
  2. Education at each follow-up visit by a specialized dietitian, reinforcing optimal diet and exercise, with pre-& post-nutrition and physical activity assessment using the validated revised summary of diabetes self-care activities (SDSCA) scale.
  3. Medication reconciliation and counseling, online post adherence questionnaire and confirm adherence by fixed medication possession ratio (FMPR) approach.
  Interventions: Other: Multifactorial intervention

INTERVENTIONS:
Other: Multifactorial intervention — 1. Correction of magnesium and/or potassium deficit and the underlying disease.
  2. Education reinforcing optimal diet and exercise, in addition to, post-nutrition assessment , diabetes self-care activities and adherence will be given at each follow up visit by a specialized dietitian.
  3. Comprehensive medication therapy management by clinical pharmacist, and medication adherence will be measured by adherence questionnaire as well as fixed medication possession ratio (FMPR).
  Arms: Multifactorial intervention group

SUMMARY:
Insufficient clinical evidence correlates the progression of diabetic kidney disease with electrolyte homeostasis in patients diagnosed with type 2 diabetes mellitus (T2DM), especially in the United Arab Emirates (UAE) population and what are the most effective interventions to slow chronic renal failure progression.

In our research, we test the hypothesis that low serum magnesium and potassium levels are directly associated with the decline of kidney function in diabetic patients who did not have severely impaired renal function at baseline. In addition, we describe the effect of long-term multifactorial adherence interventions on medication adherence, diet adherence and follow-up visits using a telemedicine approach such as mobile applications in reducing the progression of chronic kidney disease and other diabetes-related complications.

This study is a single-blind randomized control trial to demonstrate the causal relationship between potassium and magnesium levels and estimated glomerular filtration rate (eGFR) decline. The intervention group will be evaluated for manifestations of electrolyte imbalance and correction of serum magnesium and/or potassium levels will be initiated based on the last updated laboratory test. Moreover, they will receive education to reinforce diet and exercise changes at each follow up visit by a specialized dietitian with pharmacist-led comprehensive medication therapy management utilizing multifactorial adherence interventions to measure potential drug-drug or drug-food interactions, as well as medication and follow-up adherence through an integrated mobile application and fixed medication possession ratio (FMPR).

This research is under progress, and summary of its findings will be reported. This study will suggest if additional national monitoring guidelines may be warranted. In addition, it will reduce diabetic burden, medication cost in UAE and improve patient satisfaction by reducing or delaying the progression of diabetic kidney disease in diabetic patients.

DETAILED DESCRIPTION:
Some studies showed that electrolyte homeostasis is altered in diabetic patients compared with non-diabetic patients even in normotensive patients. Serum magnesium and sodium concentrations were found to be decreased and potassium and calcium levels to be increased in patients with diabetes mellitus compared to euglycemic patients (Shahid et al., 2008). Other studies showed that hyperglycemia-induced effects on cellular transport processes and the depression of the function of Sodium-potassium ATPase pump (NaK-ATPase) may play a major role in attenuating electrolyte abnormalities in patients with diabetes (Reza, et al., 2015).

Limited studies were conducted recently to investigate the effectiveness of correcting electrolyte imbalances, including both serum hypomagnesemia and hypokalemia, in improving patients' symptoms during the recovery from acute renal failure. Form several studies, the authors suggested potential avenues of future research to include investigating the effect of treating hypomagnesemia in conjunction with hypokalemia in kidney disease on the progression of diabetic kidney disease. The encouraging results of the mentioned investigation have, consequently, provoked the interest in optimizing serum magnesium and potassium to delay the progression of chronic kidney disease.

Moreover, this research will examine new dimensions of multifactorial intervention approach to the local population of UAE. The research will include dietitians' interventions to enhance adherence to dietary advice, pharmacist-led interventions to evaluate long-term adherence to medication, as well as follow-up schedule including regular laboratory testing to provide regular monitoring of eGFR, and to ensure that the patients are not receiving contraindicated or inappropriately high dose of medication as their eGFR declines in the progression of diabetic kidney.

Research Objectives The proposed research study aims to investigate the impacts of optimizing potassium and magnesium levels and multifactorial intervention including pharmacist-led medication adherence and optimization with dietary and lifestyle counseling on the progression of diabetic kidney disease and other diabetic metabolic outcomes in patients diagnosed with type 2 diabetes mellitus (T2DM) in national UAE population.

Primary Objectives:

1. To evaluate the impact on the progression of diabetic kidney disease through pharmacist-led medication compliance and optimization, along with dietary, exercise and follow-up visits adherence, using multi-intervention approach.
2. To describe the effect of pharmacist led therapy review and adherence, and dietary counseling on electrolyte levels, specifically potassium and magnesium levels.
3. To establish the relationship between serum potassium and magnesium levels and the progression of diabetic kidney disease.

Secondary objectives

1. To assess the influence of the multifactorial interventions on other diabetic outcomes, such as HbA1c level, and other diabetes-related complications.
2. To measure changes in the patient's metabolic panel and electrolyte levels as a consequence of the multifactorial interventions.

Research Overview

The proposed research will target diabetic patients and the progression of diabetic kidney disease, which is one of the most common chronic diseases among UAE citizens. The rate of progression varies considerably between individuals depending on serum electrolyte levels such as serum magnesium and potassium levels, the conventional or multifactorial intervention received, and determinants of adherence early in the course of diabetic disease. The proposed research will investigate the impact of serum magnesium and potassium levels with long-term multifactorial intervention targeting multiple risk factors and adherence on the progression of diabetic kidney disease in UAE citizen patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female UAE citizen patients between 30 and 60 years of age.
2. Patient has been previously diagnosed with type 2 diabetes mellitus recorded in Cerner, defined by diabetes mellitus in our diagnostic criteria
3. Previously on diabetic medication recorded in Cerner and antidiabetic therapy must be unchanged for 12 weeks prior to the study.
4. Patients with normal or mild to moderate magnesium and / or potassium serum levels, as defined in our definition.
5. Patients with normal or mild impaired renal function, defined as glomerular filtration rate more than 30 ml/min and albumin/creatinine ratio ≤ 30 mg/mmol, for more than 3 months as baseline value (Stage G1, G2, G3a and G3b of chronic kidney disease (CKD).
6. Body Mass index less than 40 at study enrollment.

Exclusion Criteria:

1. Non-UAE citizen patients or patients without full insurance coverage.
2. Blood dyscrasias or any disorders causing hemolysis or unstable red blood cell population (e.g., malaria, babesiosis, hemolytic anemia).
3. Patients with severe or symptomatic hypokalemia and/or hypomagnesemia, metabolic acidosis, or hypophosphatemia with or without proximal renal tubular acidosis and Fanconi syndrome, as defined in our definition.
4. Prolonged hypokalemia with surreptitious diuretic use, laxative abuse, eating disorders, or primary aldosteronism.
5. Stage 4 or 5 CKD patients, with severe reduction in glomerular filtration rate, kidney failure or dialysis, defined as GFR ≤ 29 ml/min or albumin/creatinine ratio ˃ 30 mg/mmol as baseline value.
6. High cardiovascular risk (defined as 10-year predicted ASCVD risk ≥7.5% by Pooled Cohort Equation or Framingham Risk Score ≥20%), or cardiac surgery, or angioplasty within the last 12 months or any diabetic macrovascular complications as defined in our definition.
7. Receiving medication that may cause drug-induced acute renal failure during the observational period and may be implicated in hypomagnesemia (such as aminoglycoside antibiotics, cyclosporine, amphotericin B, cisplatin, pentamidine, and foscarnet).
8. Indication of liver disease, defined by serum levels of either alanine aminotransferase (ALT), aspartate aminotransferase (AST) or alkaline phosphatase (ALP) above 3 x upper limit of normal (ULN) as determined at the beginning of the study or within the last 12 months.
9. Bariatric surgery within the past two years and other gastrointestinal surgeries that induce chronic malabsorption.
10. Medical history of cancer and/or treatment for cancer within the last 5 years, or immune compromised patients.
11. Treatment with systemic steroids or change in dosage of thyroid hormones within the last 12 months after starting the study or any other uncontrolled endocrine disorder.
12. Pre-menopausal women who are nursing or pregnant within the last 12 months.
13. Patient with communication barriers that may affect obtaining patient's adherence, receiving diet, exercise counseling or consent signing, and include:

    1. Patients with severe emotional distress.
    2. Patients who are unable to use mobile applications or to access the internet for any reason.

Ages: 30 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Difference in eGFR | From date of randomization until the end of the follow-up period or date of participant exit for any cause, whichever came first, assessed up to 12 months (during the study follow-up period)
  Difference in eGFR based on Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI) and the progression to mild albuminuria.
Serum potassium and magnesium levels | From date of randomization until the end of the follow-up period or date of participant exit for any cause, whichever came first, assessed up to 12 months (during the study follow-up period)
  The mean variation of serum potassium and magnesium levels from baseline data.
Medication adherence | From date of randomization until the end of the follow-up period or date of participant exit for any cause, whichever came first, assessed up to 12 months (during the study follow-up period)
  Change of medication adherence measured by the fixed medication possession ratio (FMPR) equation and confirmed by medication adherence questionnaire. Patient's medication refills will be recorded in each visit and the standard adherence threshold of 0.80 MPR will be used as upper bound for mediation adherence, with MPR= 1 means perfect adherence. While an MPR < 0.50 indicates patient non-adherence, and MPR=0 means no adherence.
Dietary adherence | From date of randomization until the end of the follow-up period or date of participant exit for any cause, whichever came first, assessed up to 12 months (during the study follow-up period)
  Assessment will utilize the revised Summary of Diabetes Self-Care Activities (SDSCA) scale using the metric "days per week" instead of using percentages and will cover diabetes self-care activities and adherence to the prescribed supplements during the past 7 days.
Lifestyle adherence | From date of randomization until the end of the follow-up period or date of participant exit for any cause, whichever came first, assessed up to 12 months (during the study follow-up period)
  Baseline exercise counseling by our specialized dietitian, conducted for 30 minutes at initial visit upon recruitment. Reinforcing optimal exercise level will be given at each follow up visit, with exercise post- assessment questionnaire, having 2 exercise core set questions from SDSCA scale.

SECONDARY OUTCOMES:
HbA1c level | From date of randomization until the end of the follow-up period or date of participant exit for any cause, whichever came first, assessed up to 12 months (during the study follow-up period)
  The difference in HbA1c level after one year.
Optimal electrolyte levels and metabolic panel | From date of randomization until the end of the follow-up period or date of participant exit for any cause, whichever came first, assessed up to 12 months (during the study follow-up period)
  Percentage of patients in the intervention group achieving optimal electrolyte levels and metabolic panel at the end of follow-up period.
Side effects or complications | From date of randomization until the end of the follow-up period or date of participant exit for any cause, whichever came first, assessed up to 12 months (during the study follow-up period)
  Development of any side effects or complications documented in patients' file.

CONTACTS AND LOCATIONS:
Locations (1):
- Oud Al Touba Diagnostic and Screening center, AHS, SEHA., Al Ain City, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Deyarbi M, Ahmed L, King J, Adi ZS, Al Juboori A, Mansour NA, Al Nuaimi H, Beiram R, Aburuz S. Impact of multifactorial interventions with medication and lifestyle optimization on patients with type 2 diabetes: A randomised controlled trial. PLoS One. 2025 Jul 9;20(7):e0327211. doi: 10.1371/journal.pone.0327211. eCollection 2025. PMID 40632722